CLINICAL TRIAL: NCT00005609
Title: Rituximab for Waldenstrom's Macroglobulinemia (WM): A Phase II Pilot Study for Untreated or Previously Treated Patients
Brief Title: Rituximab in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067738; E-3A98
Record Dates: First submitted 2000-05-02; First posted 2004-02-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2009-09

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Rituximab

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab in treating patients who have Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate in previously treated and previously untreated patients with Waldenstrom's macroglobulinemia receiving rituximab. II. Determine the associated toxicities with this treatment, specifically the frequency of febrile or hypotensive events, in this patient population.

OUTLINE: Patients are stratified according to prior treatment (yes vs no). Patients with prior treatment are further stratified according to type of treatment (alkylating agents vs purine nucleoside analogues). Patients receive rituximab IV over 4 hours on days 1, 8, 15, and 22. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 66 patients (33 per stratum) will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Waldenstrom's macroglobulinemia confirmed by the following: Bone marrow lymphoplasmacytosis with: Greater than 10% lymphoplasmacytic cells OR Aggregates, sheets, lymphocytes, plasma cells, or lymphoplasmacytic cells on bone marrow biopsy AND Measurable disease defined as quantitative IgM monoclonal protein greater than 1,000 mg/dL Bone marrow lymphoplasmacytosis and beta-2 microglobulin in the serum are not considered measurable Impaired bone marrow function due to infiltration by lymphoplasmacytic lymphoma Hemoglobin less than 11 g/dL OR Serum viscosity level relative to water greater than 4.0 Symptomatic with clinically significant anemia (less than 11 g/dL), bulky lymphadenopathy that is symptomatic, or symptoms attributable to hyperviscosity (e.g., nose bleeding, gingival bleeding, retinal hemorrhage)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: SGOT less than 3 times upper limit of normal Bilirubin less than 2.0 mg/dL Renal: Creatinine no greater than 3.0 mg/dL Cardiovascular: No myocardial infarction within past 6 months No significant arrhythmia within past 3 months Hypertension allowed provided controlled with medication Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Concurrent reversible complications (e.g., hyperuricemia, hyperviscosity) allowed provided therapy for complication initiated and complications subsiding Other prior malignancies allowed provided curatively treated and currently disease free

PRIOR CONCURRENT THERAPY: No more than 2 prior regimens allowed Prior tandem transplant considered 2 prior regimens Chemotherapy prior to bone marrow transplantation as part of induction considered 1 prior regimen Retreatment with same regimen (e.g., repeated alkylating agents) considered 1 prior regimen Biologic therapy: No prior anti-CD20 therapy At least 1 month since prior epoetin alfa No concurrent epoetin alfa for 2 months after registration Chemotherapy: At least 28 days since prior alkylating agents At least 28 days since prior purine nucleoside analogues Endocrine therapy: At least 28 days since prior corticosteroid therapy Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified Other: Concurrent digoxin to control atrial fibrillation allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morie A. Gertz, MD, Study Chair — Mayo Clinic
Locations (69):
- United States (66):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - Guthrie Medical Center, Sayre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Gertz MA, Abonour R, Heffner LT, Greipp PR, Uno H, Rajkumar SV. Clinical value of minor responses after 4 doses of rituximab in Waldenstrom macroglobulinaemia: a follow-up of the Eastern Cooperative Oncology Group E3A98 trial. Br J Haematol. 2009 Dec;147(5):677-80. doi: 10.1111/j.1365-2141.2009.07892.x. Epub 2009 Sep 14. PMID 19751237
- [Result] Gertz MA, Rue M, Blood E, Kaminer LS, Vesole DH, Greipp PR. Multicenter phase 2 trial of rituximab for Waldenstrom macroglobulinemia (WM): an Eastern Cooperative Oncology Group Study (E3A98). Leuk Lymphoma. 2004 Oct;45(10):2047-55. doi: 10.1080/10428190410001714043. PMID 15370249
- [Result] Ghobrial IM, Fonseca R, Greipp PR, Blood E, Rue M, Vesole DH, Gertz MA; Eastern Cooperative Oncology Group. Initial immunoglobulin M 'flare' after rituximab therapy in patients diagnosed with Waldenstrom macroglobulinemia: an Eastern Cooperative Oncology Group Study. Cancer. 2004 Dec 1;101(11):2593-8. doi: 10.1002/cncr.20658. PMID 15493038